CLINICAL TRIAL: NCT06780982
Title: The Effect of Self-care Emphasizing on Balloon-Blowing Exercise Program on Severity of Sleep Apnea and Respiratory Muscle Strength Among School Age Children With Obstructive Sleep Apnea
Acronym: "SEES"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Suwimon Rojnawee, PhD, RN, Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 829/66
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: Obstructive Sleep Apnea; Self-Efficacy; Balloon-Blowing; Muscle strength
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: The experimental group received the self-care emphasizing on balloon-blowing exercises program for five weeks based on Orem's self-care theory (2001), while the control group received regular nursing care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Balloon-blowing exercises (Experimental): The program begins with a one-on-one session on the first day of the research project and continues with home-based care through the LINE application on a smartphone for 5 weeks. The program consists of four steps:
  1. Decision-Making in Self-Care: Discussions to build rapport with the child, assess self-care deficits, and evaluate the child's current self-care behaviors based on their perceptions and experiences.
  2. Setting Goals and Planning Self-Care: Explanation self-care behaviors to the child and their parents and collaborate to create a care plan.
  3. Self-Care Implementation: The child and parents download educational materials via the LINE application and practicing the balloon-blowing exercise daily for 3 sets of 3 balloons per set (a total of 9 balloons/day), with a 1-minute rest between sets, over a period of 5 weeks.
  4. Maintaining Self-Care Behaviors: Encouragements for performing all five behaviors by having the child review materials via the LINE application once a week.
  Interventions: Behavioral: Balloon-Blowing exercise program
- Standard nursing care (Experimental): The control group received standard nursing care, which involve screening patient records and distributing educational materials in the form of brochures to individual pediatric patients and their parents. The knowledge provided in the brochures includes instructions on how to administer inhaled medication, avoiding allergens, performing facial and neck muscle exercises, and attending follow-up appointments as scheduled.
  Interventions: Behavioral: Standard nursing care

INTERVENTIONS:
Behavioral: Balloon-Blowing exercise program — he program begins with a one-on-one session on the first day of the research project and continues with home-based care through the LINE application on a smartphone for 5 weeks. The program consists of four steps:
  1. Decision-Making in Self-Care
  2. Setting Goals and Planning Self-Care
  3. Self-Care Implementation: practicing the balloon-blowing exercise daily for 3 sets of 3 balloons per set (a total of 9 balloons/day), with a 1-minute rest between sets, over a period of 5 weeks.
  4. Maintaining Self-Care Behaviors
  Arms: Experimental: Balloon-blowing exercises
Behavioral: Standard nursing care — The actions of nurses towards school-age children with obstructive sleep apnea at the hospital involve screening patient records and distributing educational materials in the form of brochures to individual pediatric patients and their parents. The knowledge provided in the brochures includes instructions on how to administer inhaled medication, avoiding allergens, performing facial and neck muscle exercises, and attending follow-up appointments as scheduled.
  Arms: Standard nursing care

SUMMARY:
Obstructive sleep apnea (OSA) is a common condition in school-age children, often leading to sleep disturbances and associated health issues. Non-invasive interventions, such as respiratory muscle training, have shown promise in mitigating the severity of OSA. This study explores the effects of a self-care-focused balloon-blowing exercise program on improving respiratory muscle strength and reducing OSA severity in children.

This research aimed to study the effects of a self-care emphasizing on balloon-blowing exercises program on severity of sleep apnea and respiratory muscle strength in school-aged children diagnosed with mild to moderate obstructive sleep apnea (OSA), receiving treatment at the outpatient ENT department at Siriraj Hospital.

DETAILED DESCRIPTION:
Thirty children participated, divided into two groups: 15 children received the self-care emphasizing on balloon-blowing exercises program for five weeks based on Orem's self-care theory (2001), and 15 children received regular nursing care. The research instruments included a severity assessment scale for apnea and a self-care behavior assessment scale for children with OSA. Both instruments had content validity indexes of 0.95 and 0.80, and their reliability, Cronbach's alpha, were 0.83 and 0.76, respectively. Respiratory muscle strength was measured using a Respiratory Pressure Meter. Data were analyzed using statistical t-tests.

ELIGIBILITY:
Inclusion Criteria:

* School-age children aged 6-12 years diagnosed with obstructive sleep apnea (OSA) of mild to moderate severity (AHI 1-9 events/hour).
* Children receiving a consistent medication dosage with no planned adjustments to increase the dosage.
* Fully conscious, with no hearing problems, and able to understand the Thai language.
* Children voluntarily agree to participate in the study, and their parents consent to provide care during the research period.
* Have a smartphone or tablet capable of using the LINE application, with the ability to operate the application under parental supervision.
* Agree to allow the researcher to communicate via LINE and phone calls.

Exclusion Criteria:

* Children with severe comorbidities or chronic illnesses requiring ongoing treatment.
* Children undergoing treatment with continuous positive airway pressure (CPAP) therapy.
* Children who have engaged in exercise sessions lasting more than 20 minutes per session, at least 3 times per week, within the 6 months prior to the start of data collection.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle strength | Change from Baseline Respiratory Muscle strength at 5 weeks
  espiratory muscle strength is assessed using a Respiratory Pressure Meter (MicroRPM®) by Micromedical, a brand from the United Kingdom. This device evaluates respiratory muscle strength by measuring the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), with results recorded in cmH₂O.
  The maximal inspiratory pressure represents the strength of the inspiratory muscles, while the maximal expiratory pressure reflects the strength of the expiratory muscles. Measurements are obtained by having the participant exert maximal and rapid respiratory effort through the Respiratory Pressure Meter, sustaining the pressure for 2 seconds. Each measurement is repeated three times, and the average of the three readings is recorded in cmH₂O.
  Higher scores indicate greater respiratory muscle strength, while lower scores signify reduced strength. The recorded data is documented in the Maximal Inspiratory and Expiratory Pressure Recording Form (Appendix D). All assessments are con

SECONDARY OUTCOMES:
Severity of sleep apnea | Change from Baseline severity of sleep apnea at 5 weeks
  The severity of sleep apnea is assessed using the Sleep-Related Breathing Disorder Pediatric Sleep Questionnaire (SRBD-PSQ), which evaluates the severity of obstructive sleep apnea (OSA). The questionnaire consists of 22 items addressing the frequency of snoring, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, hyperactivity or inattention, and symptoms of obstructive sleep apnea. Responses are scored as follows: "Yes" = 1 point, "No" = 0 points, and "Don't know" is considered missing.
  The total score is calculated by summing the scores of all answered items and dividing by the number of items answered (excluding items marked as missing). The score ranges from 0 to 1, with higher scores indicating greater severity of OSA and lower scores indicating less severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Camacho M, Certal V, Abdullatif J, Zaghi S, Ruoff CM, Capasso R, Kushida CA. Myofunctional Therapy to Treat Obstructive Sleep Apnea: A Systematic Review and Meta-analysis. Sleep. 2015 May 1;38(5):669-75. doi: 10.5665/sleep.4652. PMID 25348130
- [Result] Koka V, De Vito A, Roisman G, Petitjean M, Filograna Pignatelli GR, Padovani D, Randerath W. Orofacial Myofunctional Therapy in Obstructive Sleep Apnea Syndrome: A Pathophysiological Perspective. Medicina (Kaunas). 2021 Apr 1;57(4):323. doi: 10.3390/medicina57040323. PMID 33915707
- [Result] Schivinski CIS, Manna BC, Belem FJDM, Castilho T. THERAPEUTIC BLOWING TOYS: DOES THE OVERLAP OF VENTILATORY STIMULI ALTER THE RESPIRATORY MECHANICS OF HEALTHY SCHOOLCHILDREN? Rev Paul Pediatr. 2020 Mar 9;38:e2018259. doi: 10.1590/1984-0462/2020/38/2018259. eCollection 2020. PMID 32159645
- [Result] Zecha-Stallinger A, Wenzel V, Wagner-Berger HG, von Goedecke A, Lindner KH, Hormann C. A strategy to optimise the performance of the mouth-to-bag resuscitator using small tidal volumes: effects on lung and gastric ventilation in a bench model of an unprotected airway. Resuscitation. 2004 Apr;61(1):69-74. doi: 10.1016/j.resuscitation.2003.12.012. PMID 15081184
- [Result] Misra A, Pawar R, Pal A. Effect of Balloon-Blowing Exercise on Oxygen Saturation in COVID-19 Patients. Cureus. 2023 Jun 11;15(6):e40250. doi: 10.7759/cureus.40250. eCollection 2023 Jun. PMID 37440814
- [Result] Marcus CL, Loughlin GM. Obstructive sleep apnea in children. Semin Pediatr Neurol. 1996 Mar;3(1):23-8. doi: 10.1016/s1071-9091(96)80025-8. PMID 8795838
- [Result] Potsic WP. Sleep apnea in children. Otolaryngol Clin North Am. 1989 Jun;22(3):537-44. PMID 2657582
- [Result] Ishman SL, Li C, Dhanda Patil R. Sleep Renewed: Innovations in Sleep Apnea Care for Adults and Children. Otolaryngol Clin North Am. 2024 Jun;57(3):xv-xvi. doi: 10.1016/j.otc.2024.02.018. Epub 2024 Mar 8. No abstract available. PMID 38458954
- [Result] Redline S, Cook K, Chervin RD, Ishman S, Baldassari CM, Mitchell RB, Tapia IE, Amin R, Hassan F, Ibrahim S, Ross K, Elden LM, Kirkham EM, Zopf D, Shah J, Otteson T, Naqvi K, Owens J, Young L, Furth S, Connolly H, Clark CAC, Bakker JP, Garetz S, Radcliffe J, Taylor HG, Rosen CL, Wang R; Pediatric Adenotonsillectomy Trial for Snoring (PATS) Study Team. Adenotonsillectomy for Snoring and Mild Sleep Apnea in Children: A Randomized Clinical Trial. JAMA. 2023 Dec 5;330(21):2084-2095. doi: 10.1001/jama.2023.22114. PMID 38051326
- [Result] Erturk N, Calik-Kutukcu E, Arikan H, Savci S, Inal-Ince D, Caliskan H, Saglam M, Vardar-Yagli N, Firat H, Celik A, Yuce-Ege M, Ardic S. The effectiveness of oropharyngeal exercises compared to inspiratory muscle training in obstructive sleep apnea: A randomized controlled trial. Heart Lung. 2020 Nov-Dec;49(6):940-948. doi: 10.1016/j.hrtlng.2020.07.014. Epub 2020 Aug 13. PMID 32800391